CLINICAL TRIAL: NCT02869633
Title: Optimizing Post-allogeneic Hematopoietic Cell Transplant Outcomes for Lymphoma Using Ibrutinib
Brief Title: Ibrutinib in Treating Patients With Refractory or Relapsed Lymphoma After Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bhagirathbhai Dholaria, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC CTT 1651; NCI-2016-01246 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2016-08-10; First posted 2016-08-17 (Estimated); Results first posted 2023-01-20 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Blastoid Variant Mantle Cell Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Follicular Lymphoma; Recurrent Hodgkin Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Follicular Lymphoma; Refractory Hodgkin Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Hodgkin Disease; Lymphoma, Mantle-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ibrutinib) (Experimental): Beginning between 60-90 days post donor stem cell transplant, patients receive ibrutinib PO QD until 1 year post donor stem cell transplant in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Ibrutinib — Given by mouth
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well ibrutinib works in treating patients after a donor stem cell transplant for lymphoma that is not responding to treatment or has come back. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To study the use of ibrutinib starting between day 60 and day 90 after allogeneic hematopoietic cell transplant (HCT) until 12 months post hematopoietic cell transplant to improve the progression-free survival (PFS) at 12 months post hematopoietic cell transplant by 25% compared to historical controls.

SECONDARY OBJECTIVES:

I. To increase the incidence of successful outcome (defined as lack of requirement of second line therapy for acute graft-versus-host disease, lack of National Institutes of Health [NIH] severe chronic graft-versus-host disease, lack of progression or relapse of chronic lymphocytic leukemia/mantle cell lymphoma [MCL], lack of death from disease or non-relapse causes) to at least 60% at 1 year post hematopoietic cell transplant. (Cohort A) II. To study the safety and tolerability of ibrutinib post hematopoietic cell transplant in patients with non-Hodgkin lymphoma (NHL) and Hodgkin lymphoma. (Cohort A and B combined) III. To study the incidence of grade 3-4 acute graft-versus-host disease in the first 6 months post hematopoietic cell transplant in patients with non-Hodgkin lymphoma and Hodgkin lymphoma. (Cohort A and B combined) IV. To study the incidence of second line therapy (systemic only) for acute graft-versus-host disease in the first 6 months post hematopoietic cell transplant in patients with non-Hodgkin lymphoma and Hodgkin lymphoma. (Cohort A and B combined) V. To study the incidence of recurrent acute graft-versus-host disease in the first 6 months post hematopoietic cell transplant in patients with non-Hodgkin lymphoma and Hodgkin lymphoma. (Cohort A and B combined) VI. To study the incidence and severity of chronic graft-versus-host disease in the first 12 months post hematopoietic cell transplant in patients with not-Hodgkin lymphoma and Hodgkin lymphoma. (Cohort A and B combined) VII. To study the incidence of lung involvement with graft-versus-host disease in the first 12 months post hematopoietic cell transplant in patients with non-Hodgkin lymphoma and Hodgkin lymphoma. (Cohort A and B combined) VIII. To study the incidence of sclerotic skin chronic graft-versus-host disease in the first 12 months post hematopoietic cell transplant in patients with non-Hodgkin lymphoma and Hodgkin lymphoma. (Cohort A and B combined) IX. To study the incidence of infectious deaths not related to graft-versus-host disease in patients with non-Hodgkin and Hodgkin lymphoma. (Cohort A and B combined)

TERTIARY OBJECTIVES:

I. To study the association of minimal residual disease (MRD) as detected by immunoglobulin heavy chain (IgH) sequencing prior to starting ibrutinib and compare to post ibrutinib at month 6, 9 and 12 after HCT. (Cohort A)

II. To study the impact of onset of new acute or chronic graft-versus-host disease on minimal residual disease. (Cohort A)

III. To study the association of T-cell clonality by T cell receptor (TCR) Vb sequencing prior to starting ibrutinib and compare to post ibrutinib at month 6, 9 and 12 after hematopoietic cell transplant. (Cohort A)

IV. To study the impact of onset of new acute or chronic graft-versus-host disease on T cell receptor sequencing. (Cohort A)

V. To study the association of B cell receptor signaling pathways and immune function with response by single cell mass cytometry prior to starting ibrutinib and compare to post ibrutinib at month 6, 9 and 12 after hematopoietic cell transplant. (Cohort A)

VI. To study the association of single cell mass cytometry that investigates B cell receptor signaling and its association with new acute or chronic graft-versus-host disease on B-cell receptor (BCR) signaling. (Cohort A)

OUTLINE:

Beginning between 60-90 days post donor stem cell transplant, patients receive ibrutinib orally (PO) once daily (QD) until 1 year post donor stem cell transplant in the absence of disease progression or unacceptable toxicity.

After completion of treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

PRE-STEM CELL TRANSPLANT (SCT)

* Patients undergoing their first T cell replete allo-HCT for chronic lymphocytic leukemia (CLL), Hodgkin Lymphoma (HL), or the following subtypes of Non-Hodgkin lymphoma: Mantle cell lymphoma (MCL) and follicular center cell lymphoma (FL)
* Meeting institutional criteria for allo-HCT. Ejection fraction by echocardiogram or MUGA >40%, pulmonary function test with adjusted DLCO ≥ 60%
* Matched (8/8) or mismatched (7/8) related, unrelated HCT
* Stem cell source: bone marrow, peripheral blood stem cell
* Disease criteria:

Cohort A

Chronic lymphocytic leukemia

* Disease burden: lymph node size < 5 cm and/or extra-nodal involvement < 5 cm AND
* 17 p deletion (detected by any assay) (> or equal to 20% of cells involved if assay is conventional cytogenetics or fluorescence in situ hybridization [FISH]) or NOTCH mutation at any time point during disease course; patient should have received at least 1 line of therapy; prior ibrutinib therapy is permitted OR
* Relapsed/refractory chronic lymphocytic leukemia > or equal to 2 lines of therapy; prior ibrutinib therapy is permitted

Mantle cell lymphoma

* Disease burden: lymph node size < 5 cm and/or extra-nodal involvement < 5 cm AND
* Relapsed/refractory mantle cell lymphoma > or equal to 1 line of therapy. Prior ibrutinib therapy is permitted. Prior autologous hematopoietic cell transplant is permitted. OR
* Mantle cell lymphoma blastoid variant in first complete response (CR1) or high risk mantle cell lymphoma being considered for allo hematopoietic cell transplant in CR1

Cohort B

Follicular lymphoma

Disease burden: lymph node size < 5 cm and/or extra-nodal involvement < 5 cm AND Relapsed/refractory follicular lymphoma > or equal to 2 lines of therapy. Prior ibrutinib therapy is permitted

Hodgkin disease

* Disease burden: lymph node size < 5 cm and/or extra-nodal involvement < 5 cm AND
* Relapsed/refractory Hodgkin disease > or equal to 2 lines of therapy.

  * Preparative regimen: both reduced intensity and ablative regimens are permitted. Each center will pre-specify the regimen they intend to use during the conduct of the study
  * Donor criteria: HLA ≥ 7/8 related or unrelated donors.
  * Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
  * Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study
  * Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study
  * Prior to Administration of Ibrutinib (Day 60 to Day 90 post hematopoietic cell transplant)
* Karnofsky performance status (KPS) > or equal to 60%
* Engraftment of neutrophils (absolute neutrophil count [ANC] >= 1.0 X 10^9/L) for 3 days without granulocyte colony-stimulating factor (g-csf) support
* Platelets > or equal to 100,000/mm^3 or > or equal to = 50,000/mm^3 if bone marrow involvement independent of transfusion support in either situation
* Glomerular filtration rate (GFR) > or equal to 30 ml/min
* Liver function tests (LFTs) (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) equal to or < 3 X upper limit of normal (ULN)
* Total bilirubin equal to or < 1.5 mg/dL X ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
* Predominant donor chimerisms of > or equal to 51% as measured by CD3 and CD33 (or other myeloid marker)

Exclusion Criteria:

PRE-SCT

* Progression of chronic lymphocytic leukemia or mantle cell lymphoma or follicular lymphoma or HD at time of transplant
* Use of Coumadin (warfarin) or other vitamin-K antagonists for anticoagulation; non-Coumadin anticoagulation is permitted
* Known central nervous system involvement
* Active uncontrolled bacterial or invasive fungal infections
* History of malignancy other than the underlying disease unless treated with a curative intent and/or no evidence of disease for at least 3 years (y) OR expected to be cured with SCT
* Planned use of post-hematopoietic cell transplant cyclophosphamide for graft versus host disease prophylaxis
* Anticipated planned donor lymphocyte infusion in the first 3 months post-SCT
* T deplete hematopoietic cell transplant
* Umbilical cord hematopoietic cell transplant
* History of stroke or intracranial hemorrhage within 6 months of enrollment
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Known HIV
* Active Hepatitis B or C virus
* Child-Pugh Class C

PRIOR TO ADMINISTRATION OF IBRUTINIB (DAY 60-DAY 90 POST SCT)

* In the critical care unit, or use of mechanical ventilation or use of renal replacement therapy at any time post hematopoietic cell transplant and prior to administration of ibrutinib
* Active uncontrolled stage 3-4 acute gastrointestinal (GI) graft versus host disease prior to administration of ibrutinib
* Active uncontrolled stage 4 acute liver graft versus host disease prior to administration of ibrutinib
* Evidence of progressive disease as compared to pre-hematopoietic cell transplant (persistence of disease is permitted)
* Anticipated planned donor lymphocyte infusion in the first 3 months post-SCT
* Active uncontrolled bacterial or invasive fungal infections
* Prednisone equivalent of > 2m/kg for treatment of graft versus host disease prior to administration of ibrutinib
* Use of second line systemic therapy for treatment of acute graft versus host disease prior to administration of ibrutinib
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk. Including the presence of chronic/active HBV and HBC infections and Child-Pugh Class C.ibrutinib.
* Major surgery or a wound that has not fully healed within 4 weeks of starting.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon)
* Requires chronic treatment with strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors
* Vaccinated with live, attenuated vaccines within 4 weeks of starting ibrutinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2023-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhagirathbhai Dholaria, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (5):
- United States (5):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Stanford Cancer Institute, Palo Alto, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited participants from September 2016 through October 2019 at six medical centers.
Groups:
- Cohort A - Chronic Lymphocytic Leukemia (CLL) Mantle Cell Lymphoma (MCL); Cohort B - Follicular Lymphoma (FL) /Hodgkin Lymphoma (HL) Lymphoma (HL) Cohort: 60-90 days after donor stem cell transplant participants take Ibrutinib by mouth until 1 year after stem cell transplant.
Period: Overall Study
Arm/Group | Cohort A - Chronic Lymphocytic Leukemia (CLL) Mantle Cell Lymphoma (MCL) | Cohort B - Follicular Lymphoma (FL) /Hodgkin Lymphoma (HL) Lymphoma (HL) Cohort
Started | 16 | 7
Completed | 3 | 2
Not Completed | 13 | 5
Not completed — Death | 2 | 1
Not completed — Patient refused follow-up | 1 | 0
Not completed — Provider discretion | 1 | 0
Not completed — Investigator decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Not eligible | 6 | 1
Not completed — Protocol-defined follow-up period completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort A - CLL/MC; Cohort B - FL/HL Cohort: 60-90 days after donor stem cell transplant participants take Ibrutinib by mouth until 1 year after stem cell transplant.
- Total: Total of all reporting groups
Arm/Group | Cohort A - CLL/MC | Cohort B - FL/HL Cohort | Total
Number analyzed (Participants) | 16 | 7 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 7 | 22
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 13 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 5 | 19
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 12 | 6 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Probability at 12-month Post HCT
Description: The progression free survival (PFS) is defined as time to progression, or relapse of the underlying disease for which transplant was undertaken, or death from any non-relapse causes, starting from the date of stem cell transplant (SCT). This will be restricted to patients in cohort A which includes the diagnoses of CLL and MCL, only, and patients treated with ibrutinib. Twelve-month PFS probability with 95% confidence interval will be estimated using Kaplan-Meier method. This probability range between 0 and 1, and the higher the better.
Time Frame: Time to progression, or relapse of the underlying disease for which transplant was undertaken, or death from any non-relapse causes, assessed 12 months post HCT.
Population: Cohort A - CLL/MCL patients treated with ibrutinib starting between day 60 and day 90 after allogeneic HCT
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- Cohort A - CLL/MCL: 60-90 days after donor stem cell transplant participants take Ibrutinib by mouth until 1 year after stem cell transplant.
Arm/Group | Cohort A - CLL/MCL
Number analyzed (Participants) | 7
probability | 0.80 [0.20 to 0.97]

2. Secondary Outcome: Minimal Residual Disease Assessed by Sequencing
Time Frame: Up to 12 months
Population: Data not collected
Arm/Group | Cohort A - Chronic Lymphocytic Leukemia (CLL) Mantle Cell Lymphoma (MCL) | Cohort B - Follicular Lymphoma (FL) /Hodgkin Lymphoma (HL) Lymphoma (HL) Cohort
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: T Cell Repertoire Assessed by IMMUNOSEQ
Time Frame: Up to 12 months
Population: Data not collected
Arm/Group | Cohort A - CLL/MCL | Cohort B - FL/HL Cohort
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: B Cell Subsets and Signaling Assessed by Mass Cytometry
Time Frame: Up to 12 months
Population: Data not collected
Arm/Group | Cohort A - CLL/MCL | Cohort B - FL/HL Cohort
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: T Cell Subsets and Signaling Assessed by Mass Cytometry
Time Frame: Up to 12 months
Population: Data not collected
Arm/Group | Cohort A - CLL/MCL | Cohort B - FL/HL Cohort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Time frame for serious adverse events and other (Not Including Serious) Adverse Events: Time of consent until 30 days post cessation of study drugs up to 1 year. Time frame for All-Cause Mortality Table = Time of informed consent to off-study date, up to 2 years
Arm/Group | Cohort A - CLL/MCL | Cohort B - FL/HL Cohort
All-Cause Mortality (participants affected / at risk) | 2/16 | 1/7
Serious Adverse Events (participants affected / at risk) | 12/16 | 5/7
Other Adverse Events (participants affected / at risk) | 3/16 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - CLL/MCL (N=16) | Cohort B - FL/HL Cohort (N=7)
Febrile Neutropenia (Blood and lymphatic system disorders) | 7 (8) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3) | 0 (0)
Fever (General disorders) | 2 (3) | 3 (3)
Flu-Like Symptoms (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Altered Mental State (Psychiatric disorders) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Catheter-related Infection - MRSA (Infections and infestations) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - CLL/MCL (N=16) | Cohort B - FL/HL Cohort (N=7)
Anemia (Blood and lymphatic system disorders) | 3 (100) | 2 (2)
Platelet count decreased (Investigations) | 3 (10) | 1 (4)
Neutrophil count decreased (Investigations) | 2 (9) | 1 (1)
White blood cell decreased (Investigations) | 2 (8) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Vomitting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis, oral (Gastrointestinal disorders) | 1 (3) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Infusion-related rection (General disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT02869633/Prot_SAP_000.pdf